CLINICAL TRIAL: NCT00064636
Title: A Phase I, Open Label, Dose Escalation Study of PS-341 Plus Docetaxel in Treatment-Naive or Previously Treated Patients With Advanced Non-Small Cell Lung Cancer or Other Solid Tumors
Brief Title: Phase I Dose Escalation Study of VELCADE Plus Docetaxel in Patients With Advanced Non-Small Cell Lung Cancer or Other Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M34101-034
Record Dates: First submitted 2003-07-10; First posted 2003-07-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-09

CONDITIONS: Advanced Non-Small Cell Lung Cancer; Other Solid Tumors
MeSH Terms: interventions — Bortezomib; WW Domain-Containing Oxidoreductase

INTERVENTIONS:
Drug: VELCADE TM (bortezomib) for Injection, or PS-341

SUMMARY:
The purpose of this study is to evaluate how safe VELCADE (PS-341) is when given with Taxotere (Docetaxel) to patients with non-small cell lung cancer or other solid tumors, and also to see what effects (good and bad) it has on you and your cancer.

DETAILED DESCRIPTION:
This is a dose escalation study, which means that the first group of patients who enter the study will receive a low dose of VELCADE and Docetaxel. If the low dose of VELCADE and Docetaxel appears to be safe, then the next group of patients will receive a higher dose of VELCADE and docetaxel.

ELIGIBILITY:
Adults with advanced and/or metastatic NSCLC or other solid tumors who are treatment-naïve or previously received up to two anti-neoplastic treatment regimens and for whom there is no known curative therapy may be enrolled in this study. The actual number of patients enrolled depends on the dosing cohort in which dose-limiting toxicity is seen.

Inclusion criteria

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Patient has histologically-confirmed advanced and/or metastatic NSCLC or other solid tumors, for which the patient is treatment-naïve or previously received up to two anti-neoplastic treatment regimens and for whom there is no known curative therapy. Patients enrolled at the Low- and High- Dose Expanded Cohorts must have a diagnosis of NSCLC in order to be eligible.
* Previous treatment with carboplatin or paclitaxel does not preclude enrollment in the study.
* Patient has measurable or evaluable disease. Patients enrolled at the expanded cohorts must have measurable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines [1] presented in Table 3 and Table 4.
* Patient is 18 years of age or older.
* Patient has a Karnofsky performance status of 60% or higher.
* Patient has a life expectancy of three months or longer.
* Patient has all of the following pretreatment laboratory data within 21 days of the first study drug dose:
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mm3.
* Platelet count greater than or equal to 100,000/mm3.
* Hemoglobin greater than or equal to 8.0 g/dL.
* Serum creatinine less than or equal to 1.5 x the ULN:
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care.
* Female patient is post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) from the Screening visit through 90 days after the last study drug dose.
* Male patient agrees to use an acceptable barrier method for contraception from the Screening visit through 90 days after the last study drug dose.

Exclusion criteria

Patients meeting any of the following exclusion criteria are not to be enrolled in the study.

* Patient previously received treatment with docetaxel.
* Patient previously received treatment with cisplatin at a cumulative dose >350 mg/m2.
* Patient has received chemotherapy within four weeks, nitrosoureas within six weeks, or antibody therapy within eight weeks of enrollment.
* Patient has received radiation therapy within four weeks of enrollment.
* Patient has a history of radiation therapy to >25% of bone marrow.
* Patient has not recovered from all toxic effects of previous chemotherapy or radiation or antibody therapy.
* Patient has had any major surgery within four weeks of enrollment.
* Patient has a history of allergic reactions to appropriate diuretics or anti-emetics to be administered in conjunction with study drug.
* Patient has a history of severe hypersensitivity reaction to docetaxel or other agents formulated with polysorbate 80.
* Patient has electrocardiographic evidence of acute ischemia or new conduction system abnormalities.
* Patient has had a myocardial infarction within six months of enrollment.
* Patient has uncontrolled brain metastases or central nervous system disease.
* Patients with controlled brain metastases who are not receiving corticosteroids or anticonvulsants are eligible for study enrollment.
* Patient has Grade 2 or higher peripheral neuropathy
* Patient has leukemia or lymphoma.
* Patient has any of the following pretreatment laboratory data within 21 days before the first study drug dose:
* Total bilirubin > than the upper limit of normal (ULN).
* Alanine transaminase (ALT) and/or aspartate transaminase (AST) >1.5 x the ULN concurrent with alkaline phosphatase >2.5 x the ULN.
* Patient is HIV-infected.
* Patient is hepatitis B surface antigen positive or has previously documented hepatitis C
* Patient has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Patient has another serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Female patient is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2002-12